CLINICAL TRIAL: NCT00918723
Title: A Phase I/II Study of Fludarabine, Cyclophosphamide, Rituximab, and Vorinostat Followed by Rituximab and Vorinostat Maintenance Therapy in Patients With Previously Untreated B-Cell Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Vorinostat, Fludarabine Phosphate, Cyclophosphamide, and Rituximab in Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSOC 2401; NCI-2010-00324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PSOC 2401 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Small Lymphocytic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Small Lymphocytic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Cyclophosphamide; Rituximab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (induction and maintenance chemotherapy) (Experimental): INDUCTION THERAPY: Patients receive vorinostat PO once daily on days 1-5 and 8-12; cyclophosphamide IV over 30-60 minutes and fludarabine phosphate IV over 30-60 minutes on days 1-3; and rituximab IV on day 1, 2, 3, 4, or 5. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 3 months after the completion of induction therapy, patients receive vorinostat PO on days 1-14 and rituximab IV on day 1. Treatment repeats every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fludarabine Phosphate; Drug: Cyclophosphamide; Biological: Rituximab; Drug: Vorinostat

INTERVENTIONS:
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; SH T 586
Drug: Cyclophosphamide — Given IV
Biological: Rituximab — Given IV
  Other Names: MOAB IDEC-C2B8
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid

SUMMARY:
This phase I/II trial studies the side effects and best dose of vorinostat when given together with fludarabine phosphate, cyclophosphamide, and rituximab and to see how well they work in treating patients with previously untreated B-cell chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fludarabine phosphate and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Giving vorinostat together with fludarabine phosphate, cyclophosphamide, and rituximab may be a better treatment for CLL or SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of vorinostat that can be combined with fludarabine (fludarabine phosphate), cyclophosphamide and rituximab (FCR) in patients with previously untreated CLL/SLL.

II. To evaluate potential efficacy in terms of 2-year after FCR plus vorinostat induction followed by rituximab plus vorinostat maintenance therapy for previously untreated CLL/SLL patients.

SECONDARY OBJECTIVES:

I. To eliminate residual disease (documented by flow cytometry and/or polymerase chain reaction [PCR]) in patients who have achieved a complete response (CR) after FCR plus vorinostat.

II. To estimate the rate of conversion of partial response (PR) to CR after FCR plus vorinostat.

OUTLINE: This is a phase I, dose-escalation study of vorinostat followed by a phase II study.

INDUCTION THERAPY: Patients receive vorinostat orally (PO) once daily on days 1-5 and 8-12; cyclophosphamide intravenously (IV) over 30-60 minutes and fludarabine phosphate IV over 30-60 minutes on days 1-3; and rituximab IV on day 1, 2, 3, 4, or 5. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 3 months after the completion of induction therapy, patients receive vorinostat PO on days 1-14 and rituximab IV on day 1. Treatment repeats every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of CLL/SLL
* Patients with previously untreated cluster of differentiation (CD)20+ CLL/SLL must have either Rai stage III/IV disease or be Rai stage I/II with evidence of disease activity as defined by the National Cancer Institute (NCI) 1996 guidelines; patients with SLL must be Stage III or IV per Ann Arbor staging system
* Patient must have consented to participate in the study and signed and dated an appropriate institutional review board (IRB)-approved consent form that conforms to federal and institutional guidelines
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Patient must have an anticipated (untreated) survival of at least 3 months
* Female patient of childbearing potential has a negative serum pregnancy test beta-human chorionic gonadotropin (hCG) within 2 weeks prior to receiving the first dose of vorinostat
* Female patient is either post menopausal, free from menses for >= 2 years, surgically sterilized or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study, starting with Visit 1
* Male patients not sterilized must be willing to use adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study, starting with Visit 1
* Absolute Neutrophil Count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Prothrombin time or international normalized ratio (INR) =< 1.5 upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Partial thromboplastin time (PTT) =< 1.2 times the ULN unless the patient is receiving therapeutic anticoagulation
* Potassium level within normal limits
* Magnesium level within normal limits
* Serum creatinine =< 1.5 x ULN OR if creatinine is > 1.5 ULN the calculated creatinine clearance must be >= 60 mL/min
* Serum total bilirubin =< 1.5 times ULN; patients with Gilbert's disease or similar syndrome involving slow conjugation of bilirubin are eligible with total bilirubin > 1.5 times upper limit of normal; principal investigator (PI) review and approval required for anything above 2 times ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 ULN
* Alkaline phosphatase =< 2.5 ULN
* Patients with cytopenias due to disease or pseudohyperkalemia that do not meet these criteria, will be considered eligible with review and approval by the PI or Co-PI prior to study entry

Exclusion Criteria:

* Patients who have received cytotoxic chemotherapy, radiation therapy, immunotherapy, or cytokine treatment prior to study entry for CLL/SLL; patients who have received systemic steroids within 1 week of study entry are excluded, except patients on maintenance steroid therapy for a noncancerous disease
* Patients with active hemolysis
* Patients must not require sustained transfusion support of blood products
* Patients who have undergone treatment with either stem cell or bone marrow transplant
* Patients with active obstructive hydronephrosis
* Patients with evidence of any significant systemic illness, active hepatitis B infection, active viral hepatitis infection or other active infection at the time of study entry
* Patients with New York Heart Association class III or IV heart disease symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other serious illness, such as acute or chronic graft versus host disease, that would preclude evaluation
* Patients with congenital long QT syndrome and patients taking antiarrhythmic medicines or other medicinal products that lead to QT prolongation will only be eligible if their baseline corrected QT (QTc) prolongation is =< 500 msec
* Patients with known human immunodeficiency virus (HIV) infection
* Patients who are pregnant or nursing
* Patients with known brain or leptomeningeal involvement by malignancy
* Patients who have, in the opinion of the investigator, other medical, social, or psychosocial factors that may negatively impact compliance or their safety by participation in this study
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drugs(s)
* Patient had prior treatment with an histone deacetylases (HDAC) inhibitor (e.g., romidepsin [Depsipeptide], NSC-630176, MS 275, LAQ-824, belinostat [PXD-101], LBH589, MGCD0103, CRA024781, etc); patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* Patient with a history of a prior malignancy with the exception of cervical intraepithelial neoplasia; non-melanoma skin cancer; adequately treated localized prostate carcinoma with prostate-specific antigen (PSA) =< 1.0; or who has undergone potentially curative therapy with no evidence of that disease for five years, and/or who is deemed at low risk for recurrence by his/her treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Swedish Cancer Institute-Breast Center at First Hill Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Induction and Maintenance Chemotherapy): INDUCTION THERAPY: Patients receive vorinostat PO once daily on days 1-5 and 8-12; cyclophosphamide IV over 30-60 minutes and fludarabine phosphate IV over 30-60 minutes on days 1-3; and rituximab IV on day 1, 2, 3, 4, or 5. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Beginning 3 months after the completion of induction therapy, patients receive vorinostat PO on days 1-14 and rituximab IV on day 1. Treatment repeats every 3 months for 2 years in the absence of disease progression or unacceptable toxicity.
  Fludarabine Phosphate: Given IV
  Cyclophosphamide: Given IV
  Rituximab: Given IV
  Vorinostat: Given PO
Period: Overall Study
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 58 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32
Rai stage at the time of diagnosis [Count of Participants; unit: Participants] — Rai stage 0: Lymphocytosis in blood or bone marrow Rai stage I: Lymphocytosis + enlarged lymph nodes. Rai stage II: Lymphocytosis + enlarged liver or spleen with or without lymphadenopathy Rai stage III: Lymphocytosis + anemia (Hgb <11 g/dL) with or without enlarged liver, spleen, or lymph nodes Rai stage IV: Lymphocytosis + thrombocytopenia (platelet count <100,000/microL) with or without anemia or enlarged liver, spleen, or lymph nodes Low risk: Rai stage 0 Intermediate risk: Rai stages I and II High risk: Rai stages III and IV With higher risk, median survival outlook declines.
  Participants
    Rai stage 0 | 15
    Rai stage I/II | 19
    Rai stage III/IV | 6
Rai stage at the time of treatment [Count of Participants; unit: Participants] — Rai stage 0: Lymphocytosis in blood or bone marrow Rai stage I: Lymphocytosis + enlarged lymph nodes. Rai stage II: Lymphocytosis + enlarged liver or spleen with or without lymphadenopathy Rai stage III: Lymphocytosis + anemia (Hgb <11 g/dL) with or without enlarged liver, spleen, or lymph nodes Rai stage IV: Lymphocytosis + thrombocytopenia (platelet count <100,000/microL) with or without anemia or enlarged liver, spleen, or lymph nodes Low risk: Rai stage 0 Intermediate risk: Rai stages I and II High risk: Rai stages III and IV With higher risk, median survival outlook declines.
  Participants
    Rai stage 0 | 0
    Rai stage I/II | 23
    Rai stage III/IV | 17
Time to treatment [Mean (Full Range); unit: months] | 27 [0 to 102]
B symptoms [Count of Participants; unit: Participants] — B symptoms include weight loss, extreme fatigue, fevers, night sweats
  Participants | 13
del 17p (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 2
del 11q (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 2
Trisomy 12 (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 4
del 13q (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 3
Normal cytogenetic (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 14
Other chromosomal abnormalities (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 6
High CD38 expression (> 30%) (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 20
High ZAP-70 (> 20%) (Cytogenetics/immunophenotypic characteristics) [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat That Can be Combined With Fludarabine Phosphate, Cyclophosphamide and Rituximab (FCR) (Phase I)
Description: The MTD of vorinostat in combination with FCR will be defined as the dose level immediately below the dose level at which greater than or equal to 2 patients out of 6 of a cohort experience dose-limiting toxicity. Toxicities will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
  Doses of vorinostat analyzed to reach the MTD were 200 mg, 300 mg and 400 mg.
Time Frame: 28 days
Measure: Number; unit: mg
Groups:
- MTD for Vorinostat During Induction Therapy: MTD for patients who started induction therapy with FCR + vorinostat. Induction therapy: Patients receive vorinostat PO once daily on days 1-5 and 8-12; cyclophosphamide IV over 30-60 minutes and fludarabine phosphate IV over 30-60 minutes on days 1-3; and rituximab IV on day 1, 2, 3, 4, or 5. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  Fludarabine Phosphate: Given IV
  Cyclophosphamide: Given IV
  Rituximab: Given IV
  Vorinostat: Given PO
- MTD for Vorinostat During Maintenance Therapy: MTD for patients who started Rituximab + Vorinostat Maintenance Therapy. Maintenance therapy: Following 4-6 cycles of FCR plus vorinostat, maintenance Rituximab + Vorinostat will be given every 3 months (+/- two weeks) for 2 years. Vorinostat is given PO on days 1-14 of cycles.
  Rituximab: Given IV
  Vorinostat: Given PO
Arm/Group | MTD for Vorinostat During Induction Therapy | MTD for Vorinostat During Maintenance Therapy
Number analyzed (Participants) | 40 | 26
mg | 400 | 400

2. Primary Outcome: Percentage of Patients With Progression-free Survival at 2 Years
Description: Progression-free survival (PFS): The length of time during and after the treatment that a patient lives with the disease but it does not get worse.
  Progressive disease is specified by the NCI (National Cancer Institute) working group guidelines and additional CT (computerized tomography) scan requirements:
  Lymphadenopathy, > 50% increase in the sum of the products of at least two lymph nodes on two consecutive determinations; one lymph node must be at least 2 cm.
  An increase in the liver or spleen size by 50% or more by CT scan or the de novo appearance of hepatomegaly or splenomegaly.
  An increase in the number of blood lymphocytes by 50% or more with at least 5000 B lymphocytes per microliter.
  Transformation to a more aggressive histology or occurrence of cytopenia (neutropenia, anemia, or thrombocytopenia) attributable to CLL.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Number analyzed (Participants) | 40
percentage of participants | 87 [71 to 94]

3. Primary Outcome: Overall Survival
Description: Overall survival (OS): The percentage of people in a study who are still alive at for a certain period of time after they started treatment.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Number analyzed (Participants) | 40
percentage of participants | 90 [75 to 96]

4. Secondary Outcome: To Eliminate Residual Disease (Documented by Flow Cytometry and/or Polymerase Chain Reaction [PCR]) in Patients Who Have Achieved Complete Response (CR) After Fludarabine, Cyclophosphamide, and Rituximab (FCR) Plus Vorinostat
Time Frame: Within 21 days prior to starting maintenance therapy
Population: Patients who achieved a complete response (CR) after induction therapy and had minimal residual disease (MRD) status tested using flow cytometry
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Number analyzed (Participants) | 23
Participants
  MRD negative | 21
  MRD positive | 2

5. Secondary Outcome: To Estimate the Rate of Conversion of Partial Response (PR) to Complete Response (CR) After Fludarabine, Cyclophosphamide and Rituximab (FCR) Plus Vorinostat
Description: Responses were measured after completion of FCR+ vorinostat induction therapy (within 21 days of starting maintenance) and again after completion of maintenance therapy (24 months after the start of maintenance therapy). Maintenance therapy began within 3 months after completion of induction therapy with FCR+vorinostat. Criteria for response are specified by the National Cancer Institute (NCI) working group guidelines; in addition, patients were required to meet computed tomography (CT) criteria as described in the protocol. Response categories include Complete Response (CR), Partial Response (PR), Nodular Partial Response (nPR), Stable Disease (SD) or Progressive Disease (PD).
Time Frame: After completion of maintenance therapy (24 months after start of maintenance)
Population: Participants who had a partial response (PR) or nodular partial response (nPR) after FCR+vorinostat induction therapy, as measured within 21 days of starting maintenance therapy. Maintenance therapy began within 3 months after completion of induction therapy with FCR+vorinostat.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
Number analyzed (Participants) | 6
percentage of participants
  Conversion from PR to CR: number analyzed (Participants) | 4
  Conversion from PR to CR | 50
  Conversion from nPR (nodular PR) to CR: number analyzed (Participants) | 2
  Conversion from nPR (nodular PR) to CR | 100

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected during treatment and for 30 days after the last dose of study drug.
Arm/Group | Treatment (Induction and Maintenance Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 17/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Induction and Maintenance Chemotherapy) (N=40)
Sepsis Grade 5 (Infections and infestations) | 1 (1)
Infusion reaction Grade 3 (General disorders) | 2 (2)
Gastroenteritis Grade 3 (Gastrointestinal disorders) | 1 (1)
Dehydration Grade 3 (General disorders) | 1 (1)
Bronchiectasis Grade 3 (Infections and infestations) | 1 (1)
Sepsis Grade 4 (Infections and infestations) | 2 (2)
Diarrhea Grade 3 (Gastrointestinal disorders) | 1 (1)
Bradychardia Grade 3 (Cardiac disorders) | 1 (1)
Neutropenia Grade 3 (Blood and lymphatic system disorders) | 1 (1)
Pneumonia Grade 3 (Infections and infestations) | 1 (1)
Sepsis Grade 3 (Infections and infestations) | 1 (1)
Venous thromboemoblism Grade 4 (Vascular disorders) | 1 (1)
Drug rash with eosinophilia and systemic symptoms (DRESS) syndrome - Grade 3 (Immune system disorders) | 1 (1)
Rash Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Elective surgery (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Induction and Maintenance Chemotherapy) (N=40)
Anemia Grade 3 (Blood and lymphatic system disorders) | 2 (2)
Neutropenia Grade 2 (Blood and lymphatic system disorders) | 10 (10)
Neutropenia Grade 3 (Blood and lymphatic system disorders) | 8 (8)
Leukopenia Grade 3 (Blood and lymphatic system disorders) | 12 (12)
Neutropenia Grade 4 (Blood and lymphatic system disorders) | 16 (16)
Leukopenia Grade 4 (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia Grade 2 (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia Grade 3 (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia Grade 4 (Blood and lymphatic system disorders) | 4 (4)
Nausea Grade 3 (Gastrointestinal disorders) | 4 (4)
Vomiting Grade 3 (Gastrointestinal disorders) | 2 (2)
Constipation Grade 3 (Gastrointestinal disorders) | 2 (2)
Diarrhea Grade 3 (Gastrointestinal disorders) | 4 (4)
Gastroenteritis Grade 3 (Gastrointestinal disorders) | 1 (1)
Hyperbilirubinemia Grade 2 (Investigations) | 4 (4)
Hyperbilirubinemia Grade 3 (Investigations) | 1 (1)
Elevated alkaline phosphatase Grade 3 (Investigations) | 1 (1)
Elevated AST Grade 4 (Investigations) | 1 (1)
Elevated AST Grade 3 (Investigations) | 1 (1)
Hypoalbuminemia Grade 3 (Investigations) | 1 (1)
Elevated lipase Grade 3 (Investigations) | 1 (1)
Cholecystitis Grade 4 (Hepatobiliary disorders) | 1 (1)
Hypokalemia Grade 3 (Investigations) | 2 (2)
Hypokalemia Grade 4 (Investigations) | 1 (1)
Dehydration Grade 3 (Gastrointestinal disorders) | 1 (1)
Hypophosphatemia Grade 3 (Investigations) | 3 (3)
Renal dysfunction Grade 2 (Renal and urinary disorders) | 1 (1)
Renal dysfunction Grade 3 (Renal and urinary disorders) | 1 (1)
Hyponatremia Grade 3 (Investigations) | 1 (1)
Hypouricemia Grade 4 (Investigations) | 1 (1)
Hypocalcemia Grade 3 (Investigations) | 1 (1)
Hypertension Grade 3 (Cardiac disorders) | 1 (1)
Vasovagal episode Grade 3 (Cardiac disorders) | 1 (1)
Venous thromboembolism Grade 3 (Vascular disorders) | 2 (2)
Venous thromboembolism Grade 4 (Vascular disorders) | 1 (1)
Pneumonia Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia Grade 4 (Infections and infestations) | 1 (1)
Acute respiratory distress syndrome Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis Grade 3 (Infections and infestations) | 1 (1)
Infusion reaction Grade 2 (General disorders) | 14 (14)
Infusion reaction Grade 3 (General disorders) | 4 (4)
Infusion reaction Grade 4 (General disorders) | 1 (1)
Fatigue Grade 1 (General disorders) | 1 (1)
Fatigue Grade 3 (General disorders) | 4 (4)
Headache Grade 3 (Nervous system disorders) | 1 (1)
Back pain Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Inguinal pain Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinoma Grade 3 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rash Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
Drug rash with eosinophilia and systemic symptoms (DRESS) syndrome Grade 3 (General disorders) | 1 (1)
Hyperglycemia Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Mood alteration Grade 3 (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No